CLINICAL TRIAL: NCT03750110
Title: The Effect of Adding a Personalised Smoking Cessation Intervention to a Lung Cancer Screening Programme
Brief Title: Yorkshire Enhanced Stop Smoking Study
Acronym: YESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); University of Leeds (Other); Cardiff University (Other); University of Manchester (Other); University College, London (Other); University of York (Other); Yorkshire Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18046
Record Dates: First submitted 2018-09-17; First posted 2018-11-21 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2020-09

CONDITIONS: Cancer, Lung; Respiratory Disease; Heart Diseases
MeSH Terms: conditions — Lung Neoplasms; Respiration Disorders; Heart Diseases | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The study will use a pragmatic, parallel-group, open, randomized controlled trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Smoking Cessation NICE PH48 Guidelines
  Interventions: Other: Usual Care
- Intervention (Active Comparator): Smoking Cessation NICE PH48 Guidelines plus personalised feedback from Lung Scan
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — In addition to usual care, personalised feedback from the participants screening appointment will be provided;
  * For participants with emphysema, an image of their own emphysematous lung compared to a library image of normal lung, or a section of their own non-emphysematous lung. Where emphysema is not present, library pictures showing normal and emphysematous lung will be used.
  * For participants with coronary artery calcification, a cross sectional segment from their chest scan (either horizontal or vertical) showing the calcium compared to a library image of coronary arteries without calcification and/or a healthy section of the participant's own heart scan. Where coronary artery calcification is not present, library pictures showing normal and calcified coronary arteries will be provided.
  Arms: Intervention
Other: Usual Care — Smoking cessation support in line with NICE PH48 guidelines
  Arms: Usual Care

SUMMARY:
Lung cancer rates are higher in Yorkshire than the rest of the UK, and this is due to higher rates of smoking. Deaths from lung cancer can be reduced using regular lung scans (screening) and by helping people stop smoking. As well as detecting cancers, scans can also show evidence of damage to lungs (emphysema) and heart arteries (calcification). This study will test whether people can be encouraged to quit smoking by giving them pictures from their own scans showing possible lung and heart damage, along with information about how stopping smoking reduces their risk of cancer and heart attacks.

DETAILED DESCRIPTION:
Lung cancer has the highest mortality of all cancers in the UK and is the single biggest cause of premature death in Leeds. It disproportionately affects those from lower socioeconomically deprived communities where rates of smoking are highest. In 2014 in the Leeds South and East and the Leeds West Clinical Commissioning Group (CCG) areas, lung cancer standardized incidence rates were 131.4 and 103.3 respectively, compared to an average of 78.3 across England. Lung cancer standardized under-75 mortality rates were 52.4 and 39.3 respectively, compared to 33.26 across England. Poor outcomes from lung cancer treatment are typically the result of advanced, incurable disease at the time of symptomatic presentation. In 2011, the US National Lung Screening Trial (NLST) demonstrated a 20% reduction in lung cancer specific mortality, and a 6.7% reduction in all-cause mortality by annual low-dose CT (LDCT) screening, and lung cancer screening is now being adopted across North America having been recommended by the US Preventative Services Task Force (USPSTF) in 2013. A number of European nations are deliberating introducing screening programmes for lung cancer, and await the results of the NELSON study, the only European study powered to demonstrate a mortality reduction, which remains in follow-up. Despite widespread adoption in North America, several important questions remain regarding the best way to implement lung cancer screening. These include the optimum selection criteria to identify high-risk individuals to maximise clinical efficacy and cost-effectiveness, how to increase participation among 'hard to reach' populations, and how most effectively to embed smoking cessation support into these programmes. The Yorkshire Lung Screening Trial, funded by Yorkshire Cancer Research ( ISRCTN reference number 42704678) , seeks to address the first two issues identified above, and is due to commence screening in 2018. However, there are no currently funded UK studies specifically investigating optimal smoking cessation provision within a lung cancer screening programme.

More than 85% of cases of lung cancer are caused by tobacco smoking, and stopping smoking, at any age, significantly reduces lung cancer risk. It is therefore essential that any lung cancer screening programme provides smoking cessation support for participants, and doing so significantly increases the overall success of lung cancer screening programmes. One concern that has been raised around lung cancer screening for current smokers is the potential 'moral hazard' arising from a negative (i.e. reassuring) screening result, which may reduce motivation to quit. Conversely, attendance at a lung cancer screening programme offers a 'teachable moment' for smoking cessation, occurring at a time when participating smokers may be particularly receptive to offers of help to quit and indeed a negative screen result has been reported as being perceived as a 'clean slate' as a motivator to stop smoking. This observation fits with unpublished findings from a screening initiative in Manchester that despite a high prevalence of emphysema (68%) and coronary artery calcification (74%), most attendees were fit and relatively asymptomatic (85-90% performance status 0-1 and MRC dyspnoea scale 1-2), and hence potentially more susceptible to a message that lung damage had already occurred but clinical impact could be reduced by stopping smoking. One report from the NELSON study suggested a lower quit rate in screened persons compared to the unscreened control group, although a statistically significant effect did not persist following intention to treat analysis. No significant difference was seen between screened and control populations in the Danish Lung Cancer Screening Study, and the quit rate was significantly higher in screened versus control populations in the UK Lung Screening (UKLS) Pilot. Evidence suggests that smoking cessation and LDCT screening have additive effects on survival. An analysis of participants in the NLST reported a 38% reduction in lung cancer mortality with the combination of smoking abstinence at 15 years with LDCT screening; in addition, detection of an abnormality on the CT scan was associated with increased likelihood of smoking cessation. Further analysis of the NLST showed that arranging the smoking cessation support at the time of the screening increased quit rates by 46% (although this intervention was delivered to only 10% of study participants). In addition, research has indicated that adding smoking cessation interventions to LDCT screening improves the cost effectiveness of such programmes.

However, while smoking cessation is clearly an effective preventive intervention there is little evidence on the design and optimization of the smoking cessation interventions and support used in the screening setting. Evidence from a systematic review published in 2014 showed a benefit of materials tailored to the characteristics of individual smokers, although the included studies were conducted predominantly in the general population, rather than screening participants. Less research has been conducted investigating approaches to cessation in smokers attending for lung cancer screening, although a recent study by Marshall and colleagues reported that it was feasible to deliver a single tailored session of motivational interviewing counselling on the day of screening. For historical reasons NHS Stop Smoking Services (SSS) have evolved across the UK as opt-in facilities, whereby smokers who decide or agree to try to quit smoking then seek and are delivered help to do so. During the past five years however, evidence has grown that provision of smoking cessation support as an opt-out default generates far more quit attempts. We have demonstrated this to be the case in hospital inpatients, in which the opt-out model approximately doubled service uptake. Similar findings have been reported in relation to pregnant women setting quit dates in one NHS Foundation Trust, with uptake more than doubling after 'opt out' referrals were implemented. A study from the US found that 83% of eligible smokers did not opt out of a bedside consultation. Pro-active and systematic approaches to smoking cessation provision were recommended by NICE for pregnant women in 2010 and across all acute, maternity and mental health settings in 2013.

A recent UK study has also demonstrated the efficacy of including personalised risk information when inviting participants to smoking cessation services. A randomised controlled trial compared an individually tailored risk letter with an invitation to attend an introductory smoking cessation session to a standard generic letter advertising smoking cessation services. The personalised information was presented as a "Personal Health Risk Report", and included information on the participant's general health derived from Quality and Outcomes Framework (QOF) registered conditions on the GP record. In addition disease-specific health risks were included in the risk report, with the aim of making the individual aware of the personal health consequences of continuing to smoke, and their own individual risk of serious illness. The aim of providing this information was to change the individual's balance of perceived 'benefits' against their understanding of the harm caused by smoking. The group receiving personalised risk information had significantly higher attendance at stop smoking service (17.4% vs. 9.0%, adjusted OR 2.2, 95% CI 1.8- 2.7), higher completion of a 6-week NHS course (14.5% vs. 7.0%, adjusted OR 2.3, 95% CI 1.8-2.9) and higher 6- month validated abstinence (9.0% vs. 5.5%, adjusted OR 1.67, 95% CI 1.29-2.14).

To maximize smoking cessation among lung cancer screening participants it is therefore clearly important that all smokers who attend are provided with cessation support as a routine opt-out component of the screening visit, and that this support provides cessation pharmacotherapy and behavioural support in accordance with evidence-based NHS SSS practice. Furthermore the screening process, including risk assessment for lung cancer and imaging of the lung parenchyma and coronary arteries, allows an unprecedented opportunity for personalising the risks and harms of continued smoking, or conversely, the health gains to be made by successful smoking cessation. However there is currently no evidence on how best to design services to maximize the opportunity provided by screening participation, and how best to use the personalised information forthcoming from the screening process.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the newly merged Leeds South & East, Leeds West or Leeds North CCG
* Registered as a current or ex-smoker in a General Practice participating in YLST
* Have attended for a 'Lung Health Check' and agreed to see the SCP as part of YLST
* Smoked within the last month or have exhaled CO reading of 6ppm or above.
* Have capacity to provide informed consent.

Ages: 55 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
7-day point prevalent CO validated smoking cessation. | Three months after lung screening
  Exhaled Carbon Monoxide reading of 6ppm or less to validate smoking cessation

SECONDARY OUTCOMES:
Self-reported continuous smoking cessation at three months | Three months after lung screening
  Participant self-report being quit continuously for three months after Lung Screening. Binary question " Have you smoked in the 3 months since Lung Screening, yes or no?"
Self-reported continuous cessation at 12 months | 12 months after Lung Screening
  Participant self-reports being quit continuously for 12 months following Lung Screening. Binary question " Have you smoked in the 12 months since Lung Screening, yes or no?"
CO validated cessation at 12 months | 12 Months after lung screening
  Exhaled Carbon Monoxide reading of 6ppm or less to validate smoking cessation
Self-reported continuous cessation at 4 weeks | four weeks after lung screening
  Participant self-reports being quit continuously for 4 weeks following Lung Screening. Binary question " Have you smoked in the 4 weeks since Lung Screening, yes or no?"
CO validated cessation at 4 weeks | four weeks after lung screening
  Exhaled Carbon Monoxide reading of 6ppm or less to validate smoking cessation
Changes in perceived risk of lung cancer | 4 weeks after lung screening
  Cancer worry score (UKLS adapted version)
Changes in perceived risk of lung cancer | 3 months after lung screening
  Cancer worry score (UKLS adapted version)
Changes in perceived risk of lung cancer | 12 months after lung screening
  Cancer worry score (UKLS adapted version)
Changes in motivation to quit smoking tobacco | 12 months after lung screening
  Motivation to stop smoking - questionnaire
Changes in motivation to quit smoking tobacco | 3 months after lung screening
  Motivation to stop smoking - questionnaire
Changes in motivation to quit smoking tobacco | 4 weeks after lung screening
  Motivation to stop smoking - questionnaire
Changes in confidence and efficacy beliefs of stopping smoking | 12 months after lung screening
  Response efficacy (of stopping smoking) - questionnaire
Changes in confidence and efficacy beliefs of stopping smoking | 3 months after lung screening
  Response efficacy (of stopping smoking) - questionnaire
Changes in confidence and efficacy beliefs of stopping smoking | 4 weeks after lung health screening
  Response efficacy (of stopping smoking) - questionnaire
Confidence and efficacy beliefs of stopping smoking | 4 weeks after lung screening
  Self efficacy (of stopping smoking) - Questionnaire
Confidence and efficacy beliefs of stopping smoking | 3 months after lung screening
  Self efficacy (of stopping smoking) - Questionnaire
Confidence and efficacy beliefs of stopping smoking | 12 months after lung screening
  Self efficacy (of stopping smoking) - Questionnaire
Self -reported changes in health | 3 months after lung screening
  Health questionnaire (EQ-5D-5L)
Self -reported changes in health | 12 months after lung screening
  Health questionnaire (EQ-5D-5L)
7-day point prevalent self reported smoking cessation at 3 months | Three months after lung screening
  Exhaled Carbon Monoxide reading of 6ppm or less to validate smoking cessation

CONTACTS AND LOCATIONS:
Overall Officials: Rachael L Murray, BSc MS MSc PhD, Principal Investigator — University of Nottingham; Matthew Callister, MA, BM BCh, MEd, FRCP, PhD, Principal Investigator — The Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McInnerney D, Simmonds I, Hancock N, Rogerson S, Lindop J, Gabe R, Vulkan D, Marshall C, Crosbie PAJ, Callister MEJ, Quaife SL. Yorkshire Lung Screening Trial (YLST) pathway navigation study: a protocol for a nested randomised controlled trial to evaluate the effect of a pathway navigation intervention on lung cancer screening uptake. BMJ Open. 2024 Jul 9;14(7):e084577. doi: 10.1136/bmjopen-2024-084577. PMID 38986555
- [Derived] Murray RL, Brain K, Britton J, Quinn-Scoggins HD, Lewis S, McCutchan GM, Quaife SL, Wu Q, Ashurst A, Baldwin D, Crosbie PAJ, Neal RD, Parrott S, Rogerson S, Thorley R, Callister ME. Yorkshire Enhanced Stop Smoking (YESS) study: a protocol for a randomised controlled trial to evaluate the effect of adding a personalised smoking cessation intervention to a lung cancer screening programme. BMJ Open. 2020 Sep 10;10(9):e037086. doi: 10.1136/bmjopen-2020-037086. PMID 32912948
- [Derived] Crosbie PA, Gabe R, Simmonds I, Kennedy M, Rogerson S, Ahmed N, Baldwin DR, Booton R, Cochrane A, Darby M, Franks K, Hinde S, Janes SM, Macleod U, Messenger M, Moller H, Murray RL, Neal RD, Quaife SL, Sculpher M, Tharmanathan P, Torgerson D, Callister ME. Yorkshire Lung Screening Trial (YLST): protocol for a randomised controlled trial to evaluate invitation to community-based low-dose CT screening for lung cancer versus usual care in a targeted population at risk. BMJ Open. 2020 Sep 10;10(9):e037075. doi: 10.1136/bmjopen-2020-037075. PMID 32912947